CLINICAL TRIAL: NCT06838624
Title: Effectiveness of Treatment With RedCord in Neurogenic Bowel Dysfunction in People With Multiple Sclerosis
Brief Title: RedCord in Neurogenic Bowel Dysfunction in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Cristina Lirio, PhD, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLirio07
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis; Pelvic Floor Disorder
Keywords: Multiple Sclerosis; Constipation; Faecal Incontinence; Pelvic Floor; Abdominal Muscles
MeSH Terms: conditions — Multiple Sclerosis; Pelvic Floor Disorders; Constipation; Encopresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. It is not possible to blind the participants or the physiotherapist who will carry out the interventions; however, the researcher in charge of conducting the pre-treatment, post-treatment and follow-up assessments, and the data analyst will be blinded.
  To preserve the blindness of the evaluators and analyst, a data coding table will be used to which only the principal investigator will have access.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Redcord exercises (Experimental): The participant in this group will attend physiotherapy twice a week, every other day to avoid the onset of fatigue, for 6 weeks.
  In each physiotherapy session they will perform exercises in different plank positions using RedCord®, which is a tool with which exercises are performed in suspension and on an unstable base.
  Interventions: Device: Redcord
- Standard exercises (Active Comparator): The participant in this group will attend physiotherapy twice a week, every other day to avoid the onset of fatigue, for 6 weeks. In each physiotherapy session they will perform the same exercises as the intervention group, but on a stable basis.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Device: Redcord — Perticipants will perform exercises in different plank positions using RedCord® while applying local vibration in:
  * Supine plank position
  * Prone plank position
  * Lateral prone plank position
  Arms: Redcord exercises
Other: Control (Standard treatment) — Participants will perform exercises in different plank positions:
  Supine plank position Prone plank position Lateral prone plank position
  Arms: Standard exercises

SUMMARY:
The study aims to evaluate the effectiveness of Redcord treatment for neurogenic bowel dysfunction in patients with multiple sclerosis. The main objectives are:

* Assess the impact of Redcord on bowel function and quality of life in multiple sclerosis patients.
* Compare the outcomes of Redcord treatment with standard care practices.

Participants will undergo Redcord therapy sessions and their bowel function will be monitored and compared to a control group receiving standard care. The study will measure improvements in bowel control, frequency, and overall patient satisfaction.

DETAILED DESCRIPTION:
Study Objectives

1. Primary Objective: Assess the effectiveness of Redcord therapy in improving bowel function in MS patients.
2. Secondary Objectives:

   * To evaluate the difference in the score of the SF-36 health questionnaire and the specific quality of life questionnaire for patients with constipation CVE-20 before and after treatment, comparing these scores between the control and intervention groups.
   * To test the improvement in electrical muscle activity by electromyography of the rectus abdominis, external oblique, internal oblique, erector spinae and pelvic floor muscles and the possible relationship between the contraction of the muscles that make up the abdominal girdle (transverse abdominis, internal oblique, external oblique and rectus abdominis) and the pelvic floor muscles, comparing the control and intervention groups.

Study Design

* Type: Interventional (Clinical Trial)
* Estimated Enrollment: 76 participants
* Allocation: Randomized
* Intervention Model: Parallel Assignment
* Masking: Single (Evaluator)

Interventions

* Experimental Group: 38 participants will be randomly assigned to the intervention group who will perform exercises in different plank positions using RedCord® while applying local vibration.
* Control Group: 38 to the control group who will perform the same exercises as the intervention group, but on a stable basis.

Outcome Measures

1. Primary Outcome Measure:

   * Improvement in bowel control, measured by the Neurogenic Bowel Dysfunction Score (NBD Score) over a period of 24 weeks.

   Neurogenic Bowel Dysfunction score (NBDS) validated in Spanish is a questionnaire used for the clinical evaluation of colorectal and anal dysfunction. It is used to assess bowel dysfunction in neurological pathologies.

   It quantifies the severity of bowel dysfunction in 4 categories: very mild (score 0 to 6), mild (score 7 to 9), moderate (score 10 to 13) and severe (score greater than or equal to 14). It consists of 10 items relating to frequency of bowel movements, presence of headache and/or sweating during defecation, use of medication for constipation, time used for each defecation, frequency of bowel movements by digital extraction, frequency of faecal incontinence, medication used for faecal incontinence, presence of anal incontinence, skin problems in the peri-anal area. It also assesses the subject's satisfaction with bowel management using a score from 0 to 10, with 0 being total dissatisfaction and 10 being complete satisfaction (Cronbach's α = .97).
2. Secondary Outcome Measures:

   * Clinical data on type of multiple sclerosis, EDSS, understanding of questionnaires/surveys, pregnancy and diagnosis of severe psychological or psychiatric pathology, and demographic data on gender and age will be recorded on a questionnaire to be administered after the participant has signed the informed consent.
   * Electromyography: A Noraxon Telemyo 12-channel electromyography equipment (Noraxon USA Inc), which has been an industry leader in human movement metrics and biomechanical research for over 30 years. Electromyography data will be recorded from the rectus abdominis, external oblique, internal oblique, erector spinae and pelvic floor musculature. Rectangular, disposable, 21x41 millimetre, wireless, rectangular electrodes with gel will be used to aid electromyography. A rectal electromyographic probe will also be used to include the pelvic floor musculature.

Before placing the electrodes, the skin of each participant will be prepared. This will be done by rubbing the skin with a rough sponge, disinfecting it with isopropyl alcohol, and shaving the hair from the areas. Surface electrodes shall then be placed on the above-mentioned musculature, with an inter-electrode distance of 22 millimetres, following the direction of the muscle fibres: on the rectus abdominis the electrodes shall be aligned vertically in the centre of the muscle belly, 2 centimetres lateral and 3 centimetres superior to the umbilicus; on the external oblique they shall be placed obliquely at approximately 45° near the level of the umbilicus, midway between the rib cage and the anterior superior iliac spine; the electrodes on the internal oblique shall be placed horizontally, 2 cm inferomedial to the anterior superior iliac spine, within a triangle formed by the inguinal ligament, lateral border of the rectus sheath and the line connecting the anterior superior iliac spines; the electrodes on the erectors of the spine shall be placed 3 cm lateral to the level of L4-L5.

Water-soluble lubricant is applied to the rectal electromyography probe to facilitate intra-anal placement.

Electromyography determines muscle activity during exercise. The electrical muscle activity of the rectus abdominis, internal oblique, external oblique, spinal erectors and pelvic floor musculature will be assessed pre- and post-treatment for each participant in order to observe differences between groups using objective quantitative data. To carry out this assessment, the amplitudes of the electromyographic signals will be recorded using the Root Mean Square (RMS).

* Quality of life, assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54) questionnaire.
* Specific quality of life questionnaire for patients with constipation CVE- 20:

This is the first specific questionnaire in Spanish for patients with constipation. It is easy to complete consists of 4 dimensions: general physical, emotional, rectal physical and social. It has 5 Likert-type response options. Its scores range from 0 (worst health status) to 80 (best health status) (Cronbach's α = .87).

Eligibility Criteria

* Inclusion Criteria:
* Diagnosed with multiple sclerosis.
* Experiencing neurogenic bowel dysfunction.
* Aged 30-60 years.
* Expanded Disability Status Scale (EDSS) < 6 points.
* Able to provide informed consent.
* Exclusion Criteria:
* Severe cognitive impairment.
* Other gastrointestinal disorders.
* Pregnancy.
* Severe psychological or psychiatric pathology diagnosed.

Study Procedures

1. Screening: Eligible participants will be identified and consented.
2. Baseline Assessment: Initial evaluation of bowel function, quality of life, electromyography and other relevant parameters.
3. Intervention: Participants will undergo Redcord therapy sessions or receive standard care twice a week during 6 weeks.
4. Follow-Up Assessments: Regular monitoring of bowel function, quality of life, and patient satisfaction at 6, 12 and 24 weeks.

Data Analysis An intention-to-treat analysis will be performed. The Kolmogorov-Smirnov test will be used to determine whether a sample follows a normal distribution. All variables in this project are quantitative, therefore, they will be presented as mean ± standard deviation (SD) if they follow a parametric distribution and as median and interquartile range (IQR) if they follow a non-parametric distribution.

To analyse the relationship between the main variable and the rest of the variables investigators will use Pearson's correlation test if the data follow a normal distribution and Spearman's correlation test if the data do not follow a normal distribution.

To determine whether the intervention in the intervention group has a significant effect compared to the intervention in the control group, investigators will use the Student's t-test for independent samples if the data follow a normal distribution and the Mann-Whitney U-test if the data do not follow a normal distribution.

In assessing how the main variable changes due to the intervention, the results will be expressed as absolute differences between the initial and final measurements of the main variable.

Differences will be considered statistically significant for a p-value < 0.05. In addition, the effect size will be reported with a 95% confidence interval.

SPSS Statistics software version 29.0.2.0 will be used.

- Expected Results: It is hypothesized that Redcord therapy will significantly improve bowel function and quality of life in MS patients compared to standard care.

Ethical Considerations

* The study will be conducted in accordance with ethical principles and guidelines.
* Informed consent will be obtained from all participants.
* The study protocol will be reviewed and approved by an ethics committee.
* Researchers will undertake to comply with the ethical principles of the Declaration of Helsinki and to follow the standards of good clinical practice of the ICH (International Conference of Harmonization) Guidelines for Good Epidemiological Practice.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with Multiple Sclerosis according to McDonald's criteria.
* EDSS less than 6 points.
* Willingness to participate.

Exclusion Criteria:

* People with cognitive impairment, which makes it difficult to understand the questionnaires properly.
* Pregnant women.
* Severe psychological or psychiatric pathology diagnosed.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Neurogenic Bowel Dysfunction score (NBDS) | baseline, 6, 12 and 24 weeks
  Improvement in bowel control, measured by the Neurogenic Bowel Dysfunction Score (NBD Score) over a period of 24 weeks.
  Neurogenic Bowel Dysfunction score (NBDS) validated in Spanish is a questionnaire used for the clinical evaluation of colorectal and anal dysfunction. It is used to assess bowel dysfunction in neurological pathologies.
  It quantifies the severity of bowel dysfunction in 4 categories: very mild (score 0 to 6), mild (score 7 to 9), moderate (score 10 to 13) and severe (score greater than or equal to 14). It consists of 10 items relating to frequency of bowel movements, presence of headache and/or sweating during defecation, use of medication for constipation, time used for each defecation, frequency of bowel movements by digital extraction, frequency of faecal incontinence, medication used for faecal incontinence, presence of anal incontinence, skin problems in the peri-anal area.

SECONDARY OUTCOMES:
Electromyography: Root mean square | baseline, 6, 12 and 24 weeks
  A Noraxon Telemyo 12-channel electromyography equipment (Noraxon USA Inc). Electromyography data will be recorded from the rectus abdominis, external oblique, internal oblique, erector spinae and pelvic floor musculature. Rectangular, disposable, 21x41 millimetre, wireless, rectangular electrodes with gel will be used to aid electromyography. A rectal electromyographic probe will also be used to include the pelvic floor musculature. To carry out this assessment, the amplitudes of the electromyographic signals will be recorded using the Root Mean Square (RMS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Castilla La Macha, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No